CLINICAL TRIAL: NCT06882733
Title: The Immediate Effect of Applying Transcutaneous Electrical Nerve Stimulation (TENS) on Sympathetic Ganglion and Gastrocnemius for Popliteal Blood Flow
Acronym: TENS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Mengjie Shen, graduate student, Kaohsiung Medical University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMUHIRB-E(I)-20240357
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Transcutaneous Electrical Nerve Stimulation (TENS); Popliteal; Blood Flow; Sympathetic Ganglia
Keywords: transcutaneous electrical nerve stimulation (TENS); blood flow; sympathetic ganglia
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Sympathetic Ganglia with Low-Frequency Electrical Stimulation (Experimental): Sympathetic Ganglia (T12.L1.L2) Low-Frequency Electrical Stimulation (4Hz) electrical stimulation:15-minute
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation，TENS
- Sympathetic Ganglia with High-Frequency Electrical Stimulation (Experimental): Sympathetic Ganglia (T12.L1.L2) Low-Frequency Electrical Stimulation (80Hz) electrical stimulation:15-minute
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation，TENS
- gastrocnemius with Low-Frequency Electrical Stimulation (Experimental): gastrocnemius with Low-Frequency Electrical Stimulation Low-Frequency (4Hz) electrical stimulation:15-minute
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation，TENS
- gastrocnemius with high-Frequency Electrical Stimulation (Experimental): gastrocnemius with high-Frequency Electrical Stimulation high-Frequency(80Hz) electrical stimulation:15-minute
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation，TENS

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation，TENS — low frequency (4Hz) and sympathetic ganglion(T12.L1.L2) low frequency (4Hz) and gastrocnemius high frequency (80Hz) and sympathetic ganglion(T12.L1.L2) high frequency (80Hz) and gastrocnemius

SUMMARY:
This study aims to evaluate the immediate hemodynamic effects of transcutaneous electrical nerve stimulation (TENS) on the popliteal artery and vein. Vascular issues like PAOD and DVT are common in patients with diabetes, obesity, or immobility due to increased resistance and reduced blood flow. Traditional treatments (medication or surgery) are not always feasible, prompting interest in TENS as an alternative. Although primarily used for pain relief, TENS may enhance blood flow. This research compares different stimulation frequencies (80 Hz vs. 4 Hz) and sites (gastrocnemius muscle vs. thoracolumbar sympathetic ganglia) to identify the most effective configuration.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy people
2. Age: 18 years and above (inclusive)
3. Body mass index (BMI) between 18.5 and 24

Exclusion Criteria:

1. Unable to complete two interventions within a week
2. Have contraindications to electrotherapy (for example: metal implants in the body, open wounds, pregnancy, sensory loss)
3. Obvious varicose veins 4. Unable to lie down for about 1 to 2 hours 5. Taking drugs or nutritional supplements that affect autonomic nervous activity or vasodilation (for example: Ginkgo biloba) 6. Smoking 7. Ankle and Ankle Index (ABI) less than 0.9 or greater than 1.3

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Doppler ultrasound measurement of changes in popliteal fossa blood flow | 45 minutes
  Using Doppler ultrasound to measure blood flow before, during, immediately after, and 15 minutes after electrical stimulation to observe the effects of electrical stimulation on blood flow.

SECONDARY OUTCOMES:
heart rate | 45 minutes
  oximeter to measure heart rate before, during, immediately after, and 15 minutes after electrical stimulation to observe the effects of electrical stimulation on heart rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan, Taiwan